CLINICAL TRIAL: NCT02600624
Title: Newborn Phosphatidylethanol Screening to Detect Fetal Alcohol Exposure in Uruguay
Brief Title: Prenatal Alcohol Biomarker Study in Uruguay
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Michael Fleming, Professor in Psychiatry and Behavioral Sciences and Family and community Medicine, Northwestern University
Other Study IDs: STU00200504
Record Dates: First submitted 2015-11-03; First posted 2015-11-09 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Fetal Alcohol Syndrome
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Maternal alcohol biomarker assays will include ethylglucuronide (EtG) in hair and nails and PEth in blood obtained at the time of delivery. Newborn umbilical cord and routine 48 hour heel stick blood will be collected to assess newborn PEth levels
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants: Women who are in active labor and their newborn infants.

SUMMARY:
The purpose of this study is to examine the association between maternal alcohol use and newborn phosphatidylethanol (PEth) levels in their newborn.

DETAILED DESCRIPTION:
The goal of the proposed research study is to examine the association between maternal alcohol use and newborn phosphatidylethanol (PEth) levels in their newborn children, in a country (Uruguay) where significant alcohol use is common during pregnancy. Maternal alcohol biomarker assays will include ethyl glucuronide (EtG) in hair and nails and PEth in blood obtained at the time of delivery. Newborn umbilical cord and routine 48 hour heel stick blood will be collected to assess newborn PEth levels. Maternal biomarker levels will be compared to patient self-reported alcohol use. This proposed design is a cross-sectional study that will include 1,800 women 18 years and older and their newborns. Women who are admitted to one of two selected public health care hospitals in Montevideo, Uruguay (Hospital Pereira Rossell and Servicio Medico Integral) for obstetrical care will be recruited to participate in the study. Power estimates suggest that 1,800 maternal/infant pairs will give us sufficient power (>90%) to estimate the predictive validity of this biomarker as a routine newborn screening test.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for experimental group (n=1,800)
* Pregnant women 18 years and older
* Admitted in active labor as well as their newborn child
* Well enough to participate in the research interview
* Able to provide fingernail, hair, and blood spot samples
* All subjects must have given signed, informed consent prior to registration

Exclusion Criteria:

* Not meeting the appropriate inclusion criteria or providing consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who are admitted public health care hospitals in Montevideo, Uruguay (Hospital Pereira Rossell) for obstetrical care will be recruited to participate in the study.
Sampling Method: Probability Sample
Enrollment: 1412 (Actual)
Dates: Start 2016-08-18 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Newborn Phosphatidylethanol Screening to Detect Fetal Alcohol Exposure in Uruguay | The maternal questionnaire will occur during the 48 hrs following childbirth
  Conduct a formative assessment of the prevalence and patterns of maternal alcohol consumption during pregnancy and the relationship of these reported patterns to maternal biomarker levels (EtG in hair and nails and PEth in blood) in a large sample (n=1800) of pregnant women in Montevideo, Uruguay.

SECONDARY OUTCOMES:
Newborn Phosphatidylethanol Screening to Detect Fetal Alcohol Exposure in Uruguay | PEth and EtG Biomarkers from the mothers and newborns will be collected during the 48 hrs after childbirth.
  Biomarkers will be collected to determine the correlations between maternal self-report of alcohol consumption, maternal alcohol biomarker levels and newborn PEth concentration levels at birth. It will also help identify the sensitivity and specificity of PEth and the predictive value of newborn PEth levels; and the half-life and window of detection of PEth in newborns by examining the kinetics of PEth elimination.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fleming, MD, MPH, Principal Investigator — Northwestern University
Locations (2):
- Northwestern Memorial Hospital, Chicago, Illinois, United States
- Clínica Ginecología/Obstétrica del Hospital General de las Fuerzas Armadas de Uruguay, Montevideo, Uruguay

IPD SHARING:
Plan to Share IPD: No